CLINICAL TRIAL: NCT07366801
Title: Pilot Study of Co-Infusion of Donor Lymphocytes Enriched With Regulatory T Lymphocytes With Ex-vivo CD3-Depleted Hematopoietic Stem Cell Graft for the Prevention of Graft-versus-Host Disease in Children With Hematopoietic and Lymphoid Tissue Neoplasms
Brief Title: Co-infusion of Treg-enriched Donor Lymphocytes With CD3-depleted Hematopoietic Stem Cell Graft to Prevent Graft-versus Host Disease After Allogeneic Hematopoietic Stem Cell Transplantation Among Children With Hematologic Malignancies
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: NCHPOI- 2025-14
Record Dates: First submitted 2026-01-07; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia, Relapsed; Acute Lymphoblastic Leukemia, High Risk; Acute Myeloid Leukemia, High Risk; Acute Lymphoblastic Leukemia, Relapse
Keywords: Acute myeloid leukemia; Acute lymphoblastic leukemia; relapse; T regulatory; CD3 depletion; allogeneic HSCT
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclosporine; Sirolimus; ruxolitinib; Abatacept

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cyclosporine A (Active Comparator): Four groups corresponding to the pharmacological prophylaxis of GVHD: 1) Cyclosporine A
  Interventions: Drug: Cyclosporine A (CsA)
- Sirolimus (Active Comparator): Drug therapy (pharmacological prophylaxis of GVHD) 2) Sirolimus
  Interventions: Drug: Sirolimus
- Ruxolitinib (Active Comparator): Drug therapy (pharmacological prophylaxis of GVHD) Ruxolitinib
  Interventions: Drug: Ruxolitinib (JAKAVI®)
- Abatacept (Active Comparator): Drug therapy (pharmacological prophylaxis of GVHD) Abatacept
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Cyclosporine A (CsA) — The combination of partial T depletion and pharmacological immunosuppression minimized in volume and duration will combine the advantages of T depletion (early engraftment, low risk of GVHD, low risk of organ complications) and pharmacological prophylaxis (restoration of anti-infective immunity).
  Arms: Cyclosporine A
Drug: Sirolimus — Pharmacological prophylaxis of GVHD is one of the key subjects of evaluation in the current study. Since the optimal pharmacological approach is not known, the allocation of the patients to study groups will be by randomization procedure, although not for the purpose of direct comparison, but for unbiased descriptive analysis. There will be four main groups and an additional group to be open for allocation based on the main group closing for fitting the stopping rules. The details of pharmacological GVHD prevention are Sirolimus 1 mg -3 till +30 4-8 ng/ml
  Arms: Sirolimus
Drug: Ruxolitinib (JAKAVI®) — Pharmacological prophylaxis of GVHD is one of the key subjects of evaluation in the current study. Since the optimal pharmacological approach is not known, the allocation of the patients to study groups will be by randomization procedure, although not for the purpose of direct comparison, but for unbiased descriptive analysis. There will be four main groups and an additional group to be open for allocation based on the main group closing for fitting the stopping rules. The details of pharmacological GVHD prevention regimens are Ruxolitinib 5 mg -2 till +30
  Arms: Ruxolitinib
Drug: Abatacept — Pharmacological prophylaxis of GVHD is one of the key subjects of evaluation in the current study. Since the optimal pharmacological approach is not known, the allocation of the patients to study groups will be by randomization procedure, although not for the purpose of direct comparison, but for unbiased descriptive analysis. There will be four main groups and an additional group to be open for allocation based on the main group closing for fitting the stopping rules. Abatacept 10 mg/kg -1, +7, +14, +28
  Arms: Abatacept

SUMMARY:
Two key methods of GVHD prevention in allogeneic HSCT have a number of limitations: ex vivo T depletion is associated with an excess of infectious complications, and pharmacological immunosuppression with insufficient efficacy of GVHD prevention. Modern graft engineering technologies make it possible to create a graft with a balanced cell composition, reducing the risk of adverse events, in particular, severe forms of acute and chronic GVHD, while preserving the immunological function of the graft. In the proposed concept, enrichment of the T graft with regulatory cells will reduce the risk of GVHD and preserve a sufficient number of T lymphocytes in the graft for the formation of protective anti-infective immunity in the early stages after HSCT. The combination of partial T depletion and pharmacological immunosuppression minimized in volume and duration will combine the advantages of T depletion (early engraftment, low risk of GVHD, low risk of organ complications) and pharmacological prophylaxis (restoration of anti-infective immunity).

DETAILED DESCRIPTION:
1. Infusion of ex-vivo T-depleted peripheral blood hematopoietic stem cells (CD3 depletion product)
2. Infusion of donor lymphocytes enriched with T regulatory lymphocytes (CD25 selective product)
3. Drug therapy (pharmacological prophylaxis of GVHD)

   * Cyclosporine A
   * Sirolimus o Ruxolitinib o Abatacept

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed by the patient (age 14 to 25 years) and/or his/her legal representative (age 0 to 18 years).
2. The patient has an indication for allogeneic hematopoietic stem cell transplantation (HSCT) established in accordance with the current regulatory framework
3. Planned HSCT from a haploidentical donor
4. The Karnofsky or Lansky score is more than 70%
5. Life expectancy of at least 8 weeks
6. Heart function: ejection fraction of at least 40%
7. Consent to continue follow-up for 3 years

Exclusion Criteria:

1. Acute viral hepatitis or acute HIV infection
2. Hypoxemia with SaO2 <90%
3. Bilirubin >3 normal
4. Creatinine >3 norms
5. Pregnancy and lactation
6. Life-threatening infection
7. Severe (>?) pathology of the central nervous system (epilepsy, dementia, organic damage to the central nervous system)
8. Karnofsky score or Lansky score <70%

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-02-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility- Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | day 30
  proportion of patients who received an infusion of the planned dose of regulatory T lymphocytes (at least 80%)
Safety- Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 120 days after HSCT
  Cumulative risk of GVHD Grade III-IV (target < 5%)

SECONDARY OUTCOMES:
Cumulative probability of engraftment | up to 100 day
Time to engraftment of neutrophils and platelets | 100 day after HSCT
Cumulative risk of acute GVHD Grade II-IV | up to 100 days after HSCT
Cumulative risk of viral | at 120 day after HSCT
  (CMV, ADV, EBV, HHV-6) DNA detection in blood, peak viral DNA load and the duration of detectable viral DNA (each virus separately)
cumulative risk of developing severe chronic GVHD | at 2 years
  Severity of chronic GVHD
Cumulative risk of leukemia relapse | at 2 years
Cumulative risk of non-relapse mortality | at 100 days and 2 years
Overall survival | at 3 years
Event-free survival | at 3 years
GVHD- and relapse-free survival | at 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- National medical research center of pediatric haematology, oncology and immulogy named after Dmytriy Rogachyov, Moscow, 117198, Moscow, Russia